CLINICAL TRIAL: NCT01534299
Title: Global SYMPLICITY Registry (GSR) Denervation Findings in Real World (DEFINE)
Brief Title: Global SYMPLICITY Registry (GSR) DEFINE
Status: Recruiting | Type: Observational
Sponsor: Medtronic Vascular (Industry)
Responsible Party: Sponsor
Other Study IDs: 10031728DOC
Record Dates: First submitted 2012-02-13; First posted 2012-02-16 (Estimated); Last update posted 2025-11-26 (Actual); Status verified 2025-11

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Renal Denervation Treatment: All patients treated with renal denervation procedure will be enrolled as part of this single arm registry
  Interventions: Device: Medtronic Renal Denervation System

INTERVENTIONS:
Device: Medtronic Renal Denervation System — The Symplicity renal denervation system is comprised of a single-use, disposable catheter and a reusable radiofrequency (RF) generator. The Symplicity renal denervation system has CE Marking for the intended use of delivering low-level radiofrequency energy through the wall of the renal artery to denervate the human kidney.

SUMMARY:
This is a prospective, multi-center, single-arm, non-interventional and open-label registry. The purpose of the registry is to document the long-term safety and effectiveness of renal denervation in a real world patient population with hypertension GSR DEFINE is the continuation of the Global SYMPLICITY Registry and collectively will enroll approximately 5000 patients with hypertension who undergo the renal denervation procedure, from over 300 sites worldwide. Subjects included in GSR DEFINE will be followed for a minimum of 1 year and up to 5 years post-procedure. Patients with uncontrolled hypertension will be enrolled in accordance with the inclusion criteria specified in the protocol.

DETAILED DESCRIPTION:
This registry will collect data prospectively on patients that receive renal denervation and treatment will be applied according to the 'Intended Use' in the IFU. The treatment will be performed according to routine hospital practice and no additional tests are required specific to the registry. This registry will serve as a tool to collect clinical data in order to expand the knowledge base of safety, effectiveness and functionality of the Medtronic renal denervation system in a real world patient population.

The key measures collected for the patients will be inclusive of, but are not limited to, blood pressure measurements, change in medications, eGFR changes (based on the MDRD formula) and clinical data pertaining to hypertension .

The inclusion criteria for the registry includes:

* Age ≥ 18 years or minimum age as required by local regulations
* The patient is an acceptable candidate for renal denervation based upon the Instructions For Use for the Medtronic renal denervation system. The procedure must be performed with an initial use, market-released Medtronic renal denervation catheter.
* The patient or legal representative has been informed of the nature of the registry has consented to participate and authorized the collection and release of this medical information by signing a consent form ("Patient Informed Consent Form" or "Patient Data Release Authorization Form")

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years or minimum age as required by local regulations
* The patient is an acceptable candidate for renal denervation based upon the Instructions For Use for the Medtronic renal denervation system. The procedure must be performed with an initial use, market-released Medtronic renal denervation catheter.
* The patient or legal representative has been informed of the nature of the registry has consented to participate and authorized the collection and release of this medical information by signing a consent form ("Patient Informed Consent Form" or "Patient Data Release Authorization Form")

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects undergoing renal denervation procedure for hypertension
Sampling Method: Non-Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2012-02 (Actual); Primary Completion 2027-06 (Estimated); Study Completion 2031-12 (Estimated)

PRIMARY OUTCOMES:
BP Measurements | 6 months
  Blood pressure changes from baseline (Office Setting and 24-hr Ambulatory measurements)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Böhm, Prof., Principal Investigator — University Hospital, Saarland; Giuseppe Mancia, Prof., Principal Investigator — San Gerardo Hospital, Monza, Italy
Locations (2):
- Universitätsklinikum des Saarlandes, Homburg, Saarlandes, Germany
- Universitätsspital Basel, Basel, Switzerland

REFERENCES:
- [Derived] Nolde JM, Kiuchi MG, Carnagarin R, Ward NC, Wanten M, Bohm M, Mahfoud F, Schmieder RE, Narkiewicz K, Schlaich MP. Impact of centrally acting sympatholytic agents on the blood pressure response to renal denervation. J Hypertens. 2025 Dec 10. doi: 10.1097/HJH.0000000000004219. Online ahead of print. PMID 41411629
- [Derived] Schlaich MP, Mahfoud F, Bohm M, Narkiewicz K, Ruilope L, Williams B, Mancia G, Sharif F, Ribichini F, Lung TH, Shetty S, Schmieder RE. Renal Denervation in Patients With Moderate to Severe Chronic Kidney Disease. Hypertension. 2025 Dec;82(12):2252-2261. doi: 10.1161/HYPERTENSIONAHA.125.25470. Epub 2025 Oct 29. PMID 41159269
- [Derived] Mahfoud F, Mancia G, Schmieder RE, Ruilope L, Narkiewicz K, Schlaich M, Williams B, Ribichini F, Weil J, Almerri K, Sharif F, Lauder L, Wanten M, Fahy M, Bohm M. Outcomes Following Radiofrequency Renal Denervation According to Antihypertensive Medications: Subgroup Analysis of the Global SYMPLICITY Registry DEFINE. Hypertension. 2023 Aug;80(8):1759-1770. doi: 10.1161/HYPERTENSIONAHA.123.21283. Epub 2023 Jun 15. PMID 37317866
- [Derived] Mahfoud F, Mancia G, Schmieder RE, Ruilope L, Narkiewicz K, Schlaich M, Williams B, Ribichini F, Weil J, Kao HL, Rodriguez-Leor O, Noory E, Ong TK, Unterseeh T, de Araujo Goncalves P, Zirlik A, Almerri K, Sharif F, Lauder L, Wanten M, Fahy M, Bohm M. Cardiovascular Risk Reduction After Renal Denervation According to Time in Therapeutic Systolic Blood Pressure Range. J Am Coll Cardiol. 2022 Nov 15;80(20):1871-1880. doi: 10.1016/j.jacc.2022.08.802. PMID 36357087
- [Derived] Mahfoud F, Mancia G, Schmieder R, Narkiewicz K, Ruilope L, Schlaich M, Whitbourn R, Zirlik A, Zeller T, Stawowy P, Cohen SA, Fahy M, Bohm M. Renal Denervation in High-Risk Patients With Hypertension. J Am Coll Cardiol. 2020 Jun 16;75(23):2879-2888. doi: 10.1016/j.jacc.2020.04.036. PMID 32527396
- [Derived] Mahfoud F, Bakris G, Bhatt DL, Esler M, Ewen S, Fahy M, Kandzari D, Kario K, Mancia G, Weber M, Bohm M. Reduced blood pressure-lowering effect of catheter-based renal denervation in patients with isolated systolic hypertension: data from SYMPLICITY HTN-3 and the Global SYMPLICITY Registry. Eur Heart J. 2017 Jan 7;38(2):93-100. doi: 10.1093/eurheartj/ehw325. PMID 28158510
- [Derived] Linz D, Mancia G, Mahfoud F, Narkiewicz K, Ruilope L, Schlaich M, Kindermann I, Schmieder RE, Ewen S, Williams B, Bohm M; Global SYMPLICITY Registry Investigators. Renal artery denervation for treatment of patients with self-reported obstructive sleep apnea and resistant hypertension: results from the Global SYMPLICITY Registry. J Hypertens. 2017 Jan;35(1):148-153. doi: 10.1097/HJH.0000000000001142. PMID 27906840
- [Derived] Kim BK, Bohm M, Mahfoud F, Mancia G, Park S, Hong MK, Kim HS, Park SJ, Park CG, Seung KB, Gwon HC, Choi DJ, Ahn TH, Kim CJ, Kwon HM, Esler M, Jang YS. Renal denervation for treatment of uncontrolled hypertension in an Asian population: results from the Global SYMPLICITY Registry in South Korea (GSR Korea). J Hum Hypertens. 2016 May;30(5):315-21. doi: 10.1038/jhh.2015.77. Epub 2015 Jul 9. PMID 26155994
- [Derived] Bohm M, Mahfoud F, Ukena C, Hoppe UC, Narkiewicz K, Negoita M, Ruilope L, Schlaich MP, Schmieder RE, Whitbourn R, Williams B, Zeymer U, Zirlik A, Mancia G; GSR Investigators. First report of the Global SYMPLICITY Registry on the effect of renal artery denervation in patients with uncontrolled hypertension. Hypertension. 2015 Apr;65(4):766-74. doi: 10.1161/HYPERTENSIONAHA.114.05010. Epub 2015 Feb 17. PMID 25691618